CLINICAL TRIAL: NCT04086836
Title: Swedish Study on STroke After TAVR. A Nationwide All-comers Study of the Risk of Stroke After Transcatheter Aortic Valve Replacemant
Brief Title: Swedish Study on STroke After TAVR
Acronym: SWESTAT
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: SWESTAT
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Aortic Valve Disease; Stroke
Keywords: TAVR; Stroke
MeSH Terms: conditions — Aortic Valve Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient suffering a late stroke after TAVR: All patients suffering a stroke after TAVR will be studied
  Interventions: Device: TAVR

INTERVENTIONS:
Device: TAVR — Patient recieving a TAVR

SUMMARY:
This study aims at studying the frequency of late stroke after transcatheter aortic valve replacement/implantation

DETAILED DESCRIPTION:
Since the start of transcatheter aortic valve implnatations/replacements (TAVR/TAVI) implantations in Sweden in 2008 all procedures have been added to a national database, which now contains 5000+ procedures. At the same time, all admissions to the hospital is also recorded with diagnosis in a separate database. We intend to make a nation-wide complete follow up of all TAVR/TAVI patients in swede that has received the diagnosis of stroke after the implantation. In addition data will also be collected from the national stroke database for detailed information of the cases

ELIGIBILITY:
Inclusion Criteria:

All patients that has under TAVR/TAVI in Sweden between 2008 and 2018 Exclusion Criteria: Patients unable to follow up due to emigration or missing social security number

Exclusion Criteria:

Periprocedural stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pateints recieving a TAVR device in Sweden during study period
Sampling Method: Non-Probability Sample
Enrollment: 4600 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Stroke | 5 year
  Stroke as defined by the national stroke database

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No